CLINICAL TRIAL: NCT05153148
Title: A Phase 2b, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Multiple Dose Study to Evaluate the Efficacy, Safety, and Tolerability of NDI-034858 in Subjects With Active Psoriatic Arthritis
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of NDI-034858 in Participants With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Nimbus Lakshmi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4858-202; 2021-005888-52 (EudraCT Number)
Record Dates: First submitted 2021-11-26; First posted 2021-12-10 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Psoriatic Arthritis
Keywords: Placebo-Controlled; Double-blind; Multiple-dose study
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Treatment and randomization information will be kept confidential and will not be released to the investigator, the study staff, the contract research organization (CRO), or the sponsor's study team until after the conclusion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo capsules, orally, QD for 12 weeks.
  Interventions: Other: Placebo
- NDI-034858 Low Dose (Experimental): Participants received NDI-034858 low dose, capsules, orally, QD for 12 weeks.
  Interventions: Drug: NDI-034858
- NDI-034858 Medium Dose (Experimental): Participants received NDI-034858 medium dose, capsules, orally, QD for 12 weeks.
  Interventions: Drug: NDI-034858
- NDI-034858 High Dose (Experimental): Participants received NDI-034858 high dose, capsules, orally, QD for 12 weeks.
  Interventions: Drug: NDI-034858

INTERVENTIONS:
Drug: NDI-034858 — NDI-034858 oral capsule
  Other Names: TAK-279
  Arms: NDI-034858 High Dose; NDI-034858 Low Dose; NDI-034858 Medium Dose
Other: Placebo — NDI-034858-matching oral placebo capsule
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy, safety, and tolerability of NDI-034858 in participants with active Psoriatic Arthritis (PsA).

DETAILED DESCRIPTION:
This is a Phase 2b, Randomized, Multi-center, Double-Blind, Placebo-Controlled, Multiple Dose Study.

Randomization to one of the treatments with NDI-034858 Dose 1, 2, 3 or placebo once daily (QD) will be based on a 1:1:1:1 scheme.

The maximum study duration per participant is approximately 20 weeks, including up to 30 days for the screening period, a 12-week treatment period, and a 4-week safety follow-up period.

Efficacy will be assessed using the ACR20 composite measure (including tender and swollen joint count, patient assessment of PsA pain visual analog scale (VAS), patient global PsA assessment VAS, physician global PsA assessment, HAQ-DI, and hsCRP) as well as the additional components. Efficacy for psoriasis among participants who have ≥ 3% BSA) involvement on Day 1, will be measured using PASI, PGAs, and BSA.

Safety will be assessed by collecting AEs, recording vital signs, performing physical examinations, and evaluating clinical laboratory and ECGs results.

Blood samples will be collected to measure plasma concentrations of NDI-034858.

ELIGIBILITY:
Inclusion Criteria:

* Participant has PsA on the basis of the Classification Criteria for Psoriatic Arthritis with peripheral symptoms at the screening visit.
* Participant has a history of PsA symptoms for ≥ 6 months prior to the screening visit.
* Participant has ≥ 3 tender joints and ≥ 3 swollen joints at screening and Day 1 visits.
* Participant has at least one lesion of plaque psoriasis ≥ 2 cm in diameter, nail changes characteristic of psoriasis, or a documented history of plaque psoriasis.
* Participant has active PsA despite previous standard doses of non-steroidal anti-inflammatory drug (NSAIDs) administered for ≥ 4 weeks, or traditional disease-modifying anti-rheumatic drug (DMARDs) (including methotrexate and sulfasalazine) administered for ≥ 3 months, or tumor necrosis factor inhibitor (TNFi) agents administered for ≥ 3 months, or participants are intolerant to NSAIDs or DMARDs or TNFi agents.
* If participant is on concurrent PsA treatments, they must be on stable doses.
* All female participants should followed the protocol defined contraceptive method.

Exclusion Criteria:

* Participant has other disease(s) that might confound the evaluations of benefit of NDI-034858 therapy, including but not limited to rheumatoid arthritis (RA), axial spondyloarthritis (this does not include a primary diagnosis of PsA with spondylitis), systemic lupus erythematosus, Lyme disease, or fibromyalgia.
* Participant has a history of lack of response to any therapeutic agent targeting IL-12, IL17, and/or IL23 at approved doses after at least 12 weeks of therapy, and/or received one of these therapies within 6 months prior to baseline (Day 1).
* Participant has a history of lack of response to > 1 therapeutic agent targeting tumor necrosis factor.
* Participant has received infliximab, golimumab, adalimumab, or certolizumab pegol, or any biosimilar of these agents, within 8 weeks prior to baseline (Day 1).
* Participant has received etanercept, or any biosimilar of etanercept, within 4 weeks prior to baseline (Day 1).
* Participant has received rituximab or any immune-cell-depleting therapy within 6 months prior to baseline (Day 1).
* Participant has received any marketed or investigational biological agent, other than those specified in other inclusion/exclusion criteria, within 12 weeks or 5 half-lives prior to baseline (Day 1).
* Participant is currently receiving a non-biological investigational product or device or has received one within 4 weeks prior to baseline (Day 1).
* Participant has received apremilast or other non-biologic systemic treatment for PsA within 4 weeks prior to baseline (Day 1), other than methotrexate (MTX), sulfasalazine, corticosteroids, NSAIDs, or paracetamol/acetaminophen, which are allowed at stable doses as described in Inclusion Criterion 7. For participants not receiving MTX and sulfasalazine at screening, MTX and sulfasalazine are excluded within 4 weeks prior to baseline (Day 1). Participant has received leflunomide within 8 weeks of baseline (Day 1) if no elimination procedure was followed or adhere to an elimination procedure. For participants not receiving MTX and sulfasalazine at Screening, MTX and sulfasalazine are excluded within 4 weeks prior to baseline (Day 1).
* Participant has received intraarticular injection (including corticosteroids), intramuscular steroids, intralesional steroids, or intravenous steroids within 4 weeks prior to baseline (Day 1). For participants not receiving MTX and sulfasalazine at screening, MTX and sulfasalazine are excluded within 4 weeks prior to baseline (Day 1). For participants not receiving MTX and sulfasalazine at screening, MTX and sulfasalazine are excluded within 4 weeks prior to baseline (Day 1).
* Participant has received high potency opioid analgesics (eg, methadone, hydromorphone, or morphine) within 2 weeks prior to baseline (Day 1).
* Participant has used any topical medication that could affect PsA or psoriasis (including corticosteroids, retinoids, vitamin D analogues (such as calcipotriol), JAK inhibitors, or tar) within 2 weeks prior to baseline (Day 1).
* Participant has used any systemic treatment that could affect PsA or psoriasis (including oral retinoids, immunosuppressive/immunomodulating medication, cyclosporine, oral JAK inhibitors, or apremilast) within 4 weeks prior to baseline (Day 1).
* Participant has received any ultraviolet (UV)-B phototherapy (including tanning beds) or excimer laser within 4 weeks prior to baseline (Day 1).
* Participant has had psoralen and UV A (PUVA) treatment within 4 weeks prior to baseline (Day 1).
* Participant has received Chinese traditional medicine within 4 weeks prior to baseline (Day 1)
* Participant has received any live-attenuated vaccine, including for COVID-19, within 4 weeks prior to baseline (Day 1) or plans to receive a live-attenuated vaccine during the study and up to 4 weeks or 5 half-lives of the study drug, whichever is longer, after the last study drug administration.
* Participant is currently being treated with strong or moderate cytochrome P450 3A (CYP3A4) inhibitors, such as itraconazole or has received moderate or strong CYP3A4 inhibitors within 4 weeks prior to baseline (Day 1).
* Participant has consumed grapefruit or grapefruit juice within 1 week prior to baseline (Day 1).
* Participant has used tanning booths within 4 weeks prior to baseline (Day 1), has had excessive sun exposure, or is not willing to minimize natural and artificial sunlight exposure during the study.
* Participant is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
* Participant has evidence of erythrodermic, pustular, predominantly guttate psoriasis, or drug-induced psoriasis.
* Participant has any clinically significant medical condition, evidence of an unstable clinical condition, psychiatric condition, or vital signs/physical/laboratory/ECG abnormality that would, in the opinion of the investigator, put the participant at undue risk or interfere with interpretation of study results.
* Participant had a major surgery within 8 weeks prior to baseline (Day 1 or has a major surgery planned during the study.
* Participant has a history of Class III or IV congestive heart failure as defined by New York Heart Association Criteria.
* Participant has an estimated creatinine clearance of < 40 mL/min based on the Cockcroft-Gault equation or a history of renal failure.
* Participant was hospitalized in the 3 months prior to screening for asthma, has ever required intubation for treatment of asthma, currently require oral corticosteroids for the treatment of asthma, or has required more than one short-term (≤ 2 weeks) course of oral corticosteroids for asthma within 6 months prior to baseline (Day 1).
* Participant has a history of cancer or lymphoproliferative disease within 5 years prior to baseline (Day 1). Participants with successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded.
* Participant has a history of fever, inflammation, or systemic signs of illness suggestive of systemic or invasive infection within 4 weeks prior to baseline (Day 1).
* Participant has an active bacterial, viral, fungal, mycobacterial infection, or other infection (including TB or atypical mycobacterial disease), or any major episode of infection that required hospitalization or treatment with intravenous antibiotics within 12 weeks prior to baseline (Day 1), or oral antibiotics within 4 weeks prior to baseline (Day 1).
* Participant has a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection, recurrent urinary tract infection, fungal infection (with the exception of superficial fungal infection of the nailbed), or infected skin wounds or ulcers.
* Participant has a history of an infected joint prosthesis or has received antibiotics for a suspected infection of a joint prosthesis, if that prosthesis has not been removed or replaced.
* Participant has active herpes infection, including herpes simplex 1 and 2 and herpes zoster within 8 weeks prior to Day 1.
* Participant has a history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the Participant's immune status (eg, history of splenectomy, primary immunodeficiency).
* Participant has positive results for hepatitis B surface antigens (HBsAg), antibodies to hepatitis B core antigens (anti-HBc), hepatitis C virus (HCV), or human immunodeficiency virus (HIV). Samples testing positive for HCV antibodies will require polymerase chain reaction (PCR) qualitative testing for HCV RNA.
* Participant has clinical or laboratory evidence of active or latent TB infection at screening as assessed by QuantiFERON-TB Gold (or a purified protein derivative [PPD] skin test or equivalent, or both if required per local guidelines) and chest X-ray. The PPD skin test should be utilized only when a QuantiFERON-TB Gold Test is not possible for any reason (unless local guidelines require both tests). Chest X-ray may be taken at screening or completed within 3 months prior to the screening visit, with documentation showing no evidence of infection or malignancy as read by a qualified physician.
* Participant has a known or suspected allergy to NDI-034858 or any component of the investigational product, or any other significant drug allergy (such as anaphylaxis or hepatotoxicity).
* Participant has a known history of clinically significant drug or alcohol abuse in the last year prior to baseline (Day 1).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (48):
- United States (22):
  - Nimbus site #XYZ, Palm Desert, California
  - Nimbus site #XYZ, Upland, California
  - Nimbus site #XYZ, Hollywood, Florida
  - Nimbus site #XYZ, Plantation, Florida
  - Nimbus site #XYZ, St. Petersburg, Florida
  - Nimbus site #XYZ, Tampa, Florida
  - Nimbus site #XYZ, Winter Park, Florida
  - Nimbus site #XYZ, Zephyrhills, Florida
  - Nimbus site #XYZ, Indianapolis, Indiana
  - Nimbus site #XYZ, West Des Moines, Iowa
  - Nimbus site #XYZ, Lake Charles, Louisiana
  - Nimbus site #XYZ, Worcester, Massachusetts
  - Nimbus site #XYZ, Albuquerque, New Mexico
  - Nimbus site #XYZ, Charlotte, North Carolina
  - Nimbus site #XYZ, Duncansville, Pennsylvania
  - Nimbus site #XYZ, Columbia, South Carolina
  - Nimbus site #XYZ, Jackson, Tennessee
  - Nimbus site #XYZ, Baytown, Texas
  - Nimbus site #XYZ, Corpus Christi, Texas
  - Nimbus site #XYZ, Houston, Texas
  - Nimbus site #XYZ, Mesquite, Texas
  - Nimbus site #XYZ, Beckley, West Virginia
- Czechia (6):
  - Nimbus site #XYZ, Hlučín, Ostrava-město
  - Nimbus site #XYZ, Prague, Praha 3
  - Nimbus site #XYZ, Ostrava
  - Nimbus site #XYZ, Pardubice
  - Nimbus site #XYZ, Uherské Hradiště
  - Nimbus site #XYZ, Zlín
- Germany (7):
  - Nimbus site #XYZ, Cottbus, Brandenburg
  - Nimbus site #XYZ, Bonn, North Rhine-Westphalia
  - Nimbus site #XYZ, Cologne, North Rhine-Westphalia
  - Nimbus site #XYZ, Herne, North Rhine-Westphalia
  - Nimbus site #XYZ, Ratingen, North Rhine-Westphalia
  - Nimbus site #XYZ, Berlin
  - Nimbus site #XYZ, Hamburg
- Poland (13):
  - Nimbus site #XYZ, Krakow, Lesser Poland Voivodeship
  - Nimbus site #XYZ, Lublin, Lublin Voivodeship
  - Nimbus site #XYZ, Elblag, Warmian-Masurian Voivodeship
  - Nimbus site #XYZ, Bialystok
  - Nimbus site #XYZ, Bydgoszcz
  - Nimbus site #XYZ, Krakow
  - Nimbus site #XYZ, Nadarzyn
  - Nimbus site #XYZ, Nowa Sól
  - Nimbus site #XYZ, Poznan
  - Nimbus site #XYZ, Sochaczew
  - Nimbus site #XYZ, Torun
  - Nimbus site #XYZ, Warsaw
  - Nimbus site #XYZ, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/dcef5a65f54b4529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 45 investigative sites in the United States (US), Germany, Poland, and the Czech Republic from 6 January 2022 to 2 June 2023.
Pre-assignment Details: A total of 305 participants with a diagnosis of psoriatic arthritis were enrolled in a 1:1:1:1 ratio to receive either one of the 3 doses of NDI-034858 or placebo.
Groups:
- Placebo: Participants received placebo capsules, orally, once daily (QD) for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Started | 75 | 76 | 78 | 76
Completed | 66 | 66 | 65 | 60
Not Completed | 9 | 10 | 13 | 16
Not completed — Adverse Event | 1 | 0 | 3 | 5
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 6 | 8 | 6 | 8
Not completed — Coronavirus Disease 2019 (COVID-19) | 0 | 0 | 1 | 0
Not completed — Randomized Without Dosing due to Ineligibility | 0 | 0 | 0 | 2
Not completed — Reason not Specified | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose | Total
Number analyzed (Participants) | 72 | 71 | 75 | 72 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (11.83) | 48.3 (10.43) | 52.5 (12.15) | 49.0 (11.51) | 49.9 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 40 | 46 | 43 | 166
  Male | 35 | 31 | 29 | 29 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 4 | 2 | 9
  Not Hispanic or Latino | 70 | 69 | 71 | 70 | 280
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69 | 66 | 71 | 69 | 275
  Non-white | 1 | 3 | 4 | 3 | 11
  Missing | 2 | 2 | 0 | 0 | 4
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 170.3 (10.65) | 170.1 (8.67) | 169.0 (9.04) | 170.4 (9.06) | 169.9 (9.35)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 86.26 (25.307) | 86.97 (26.611) | 85.85 (22.048) | 87.74 (20.152) | 86.69 (23.529)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI = weight (kg)/[height (m)^2]
  kilograms per meter square (kg/m^2) | 29.48 (6.865) | 29.78 (8.153) | 30.04 (7.937) | 30.15 (6.610) | 29.87 (7.390)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved at Least an American College of Rheumatology 20 (ACR20) Response at Week 12
Description: ACR20 is composite measure defined as improvement of 20 percent(%) from baseline in both number of tender (68) & number of swollen (66) joints & a 20% improvement in at least 3 of following 5 criteria: patient global assessment of psoriatic arthritis (PGA-PsA) [visual analog scale (VAS) where, 0=very good, no symptoms & 100=very poor, severe symptoms], physician global assessment of psoriatic arthritis (PhGA-PsA) [(VAS) where 0=no disease activity & 100=maximum disease activity], patient global assessment of psoriatic arthritis pain (PGAAP) [(VAS) where 0=no pain & 100=most severe pain], disability history questionnaire i.e., Health Assessment Questionnaire-Disability Index [HAQ-DI] (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip & activities, 0=without difficulty to 3=unable to do) & acute phase reactant like high sensitivity C-reactive protein [hsCRP]). Percentages are rounded off to the nearest decimal.
Time Frame: Week 12
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 72 | 71 | 75 | 72
percentage of participants | 29.2 [18.7 to 39.7] | 35.2 [24.1 to 46.3] | 53.3 [42.0 to 64.6] | 54.2 [42.7 to 65.7]
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.446, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.9, 95% CI 2-sided [-9.3 to 21.1] — Mantel-Haenszel (MH) risk difference was summarized along with the 2-sided 95% confidence interval (CI) using MH stratum weights and the Sato variance estimator; Comparisons of ACR20 responder rates at Week 12 were made independently between each dose group and the placebo group using two-sided MH tests stratified on randomization stratification factors: prior treatment with biologics or non-traditional disease-modifying antirheumatic drugs (DMARDs) and region
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.1, 95% CI 2-sided [8.6 to 39.6] — MH risk difference was summarized along with the 2-sided 95% CI using MH stratum weights and the Sato variance estimator; Comparisons of ACR20 responder rates at Week 12 were made independently between each dose group and the placebo group using two-sided MH tests stratified on randomization stratification factors: prior treatment with biologics or non-traditional DMARDs and region
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.5, 95% CI 2-sided [9.0 to 39.9] — [estimate comment as in outcome 1, analysis 2]; [other analysis details as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants Who Achieved at Least an ACR-50 Response at Week 12
Description: The ACR-50 is a composite measure defined as improvement of 50% from baseline in both the number of tender (68) and number of swollen (66) joints, and a 50% improvement in at least three of the following five criteria: PGA-PsA (VAS where, 0 is 'very good, no symptoms' and 100 is 'very poor, severe symptoms'), PhGA-PsA [(VAS) where 0=no disease activity and 100=maximum disease activity], PGAAP [(VAS) where 0=no pain & 100=most severe pain], disability history questionnaire (i.e., HAQ-DI) [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do] and an acute phase reactant [i.e., erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)]. Percentages are rounded off to the nearest decimal.
Time Frame: Week 12
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 72 | 71 | 75 | 72
percentage of participants | 9.7 [2.9 to 16.6] | 15.5 [7.1 to 23.9] | 26.7 [16.7 to 36.7] | 26.4 [16.2 to 36.6]
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.312, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.7, 95% CI 2-sided [-5.3 to 16.6] — [estimate comment as in outcome 1, analysis 2]; Comparisons of ACR50 responder rates at Week 12 were made independently between each dose group and the placebo group using two-sided MH tests stratified on randomization stratification factors: prior treatment with biologics or non-traditional DMARDs and region
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.0, 95% CI 2-sided [5.0 to 29.1] — [estimate comment as in outcome 1, analysis 2]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.4, 95% CI 2-sided [4.2 to 28.6] — [estimate comment as in outcome 1, analysis 2]; [other analysis details as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants Who Achieved at Least an ACR-70 Response at Week 12
Description: The ACR-70 is a composite measure defined as improvement of 70% from baseline in both the number of tender (68) and number of swollen (66) joints, and a 70% improvement in at least three of the following five criteria: PGA-PsA (VAS where, 0 is 'very good, no symptoms' and 100 is 'very poor, severe symptoms'), PhGA-PsA [(VAS) where 0=no disease activity and 100=maximum disease activity], PGAAP [(VAS) where 0=no pain & 100=most severe pain], disability history questionnaire (i.e., HAQ-DI) [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do] and an acute phase reactant (i.e., ESR or CRP). Percentages are rounded off to the nearest decimal.
Time Frame: Week 12
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 72 | 71 | 75 | 72
percentage of participants | 5.6 [1.5 to 13.6] | 8.5 [2.0 to 14.9] | 14.7 [6.7 to 22.7] | 13.9 [5.9 to 21.9]
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.532, Fisher Exact; Risk Difference (RD) = 2.9, 95% CI 2-sided [-6.6 to 12.7] — Comparisons of ACR70 responder rates at Week 12 were made independently between each dose group and the placebo group using Fischer's exact Method
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.101, Fisher Exact; Risk Difference (RD) = 9.1, 95% CI 2-sided [-1.0 to 20.1] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.158, Fisher Exact; Risk Difference (RD) = 8.3, 95% CI 2-sided [-1.7 to 19.4] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Week 12
Description: The TJC 68 is a total score of points assigned for the presence of tenderness in the 68 joints in the upper body and upper/lower extremity. The response to tenderness for each joint was evaluated using the following scale: 'Present' was assigned a score of 1 whereas, 'Absent', 'Not Done', 'Not Applicable', or joints with missing response were assigned a score of 0. The sum of all tender joints was derived. The overall tender joint count ranged from 0 to 68, with a higher score indicating a greater degree of tenderness. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug. Overall number analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: tender joints
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 66 | 66 | 64 | 63
tender joints | -5.9 (1.12) | -7.6 (1.12) | -8.9 (1.12) | -8.3 (1.15)
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.268, Mixed Model Repeated Measure (MMRM); Treatment Difference = -1.7, 95% CI 2-sided [-4.8 to 1.3] — Point estimate and 95% CI were obtained from a MMRM model; MMRM model included fixed effects for treatment group, visit, and treatment group-by-visit interaction, with baseline value and the randomization stratification factors (prior treatment with biologics or non-traditional DMARDs and region) as covariates, and the change from baseline as the dependent variable
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.051, MMRM; Treatment Difference = -3.0, 95% CI 2-sided [-6.1 to 0.0] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.112, MMRM; Treatment Difference = -2.5, 95% CI 2-sided [-5.6 to 0.6] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Week 12
Description: The SJC 66 (TJC 68 joint assessment minus hip joints, which cannot be assessed for swelling) is a total score of points assigned for presence of swelling in the 66 joints in the upper body and upper/lower extremity. The response to swelling for each joint was evaluated using the following scale: 'Present' was assigned a score of 1 whereas, 'Absent', 'Not Done', 'Not Applicable', or joints with missing response were assigned a score of 0. The sum of all swollen joints was derived. The overall swollen joint count ranged from 0 to 66, with a higher score indicating a greater degree of swelling. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 66 | 66 | 64 | 63
swollen joints | -3.9 (0.57) | -4.8 (0.58) | -5.0 (0.58) | -5.0 (0.59)
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.280, MMRM; Treatment Difference = -0.9, 95% CI 2-sided [-2.4 to 0.7] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.177, MMRM; Treatment Difference = -1.1, 95% CI 2-sided [-2.6 to 0.5] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.196, MMRM; Treatment Difference = -1.0, 95% CI 2-sided [-2.6 to 0.5] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: Change From Baseline in PGA-PsA at Week 12
Description: Participants assessed their overall disease status based on symptoms of psoriasis and psoriatic arthritis at the time of the visit using the PGA-PsA VAS of 100 millimeters (mm) which ranges from 0 (very good, no symptoms) to 100 (very poor, severe symptoms). A negative change from Baseline indicates improvement in symptoms.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 64 | 65 | 63 | 62
mm | -11.1 (2.85) | -12.9 (2.84) | -20.2 (2.85) | -19.8 (2.92)
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.637, MMRM; Treatment Difference = -1.9, 95% CI 2-sided [-9.6 to 5.9] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.021, MMRM; Treatment Difference = -9.2, 95% CI 2-sided [-17.0 to -1.4] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.030, MMRM; Treatment Difference = -8.7, 95% CI 2-sided [-16.5 to -0.9] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]

7. Secondary Outcome: Change From Baseline in PGAAP at Week 12
Description: Participants assessed their overall psoriatic arthritis-related pain at the time of the visit using the PGAAP VAS of 100 mm which ranges from 0 (no pain) to 100 (most severe pain). A negative change from Baseline indicates improvement in pain.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 64 | 65 | 63 | 62
mm | -12.1 (2.75) | -13.0 (2.74) | -18.8 (2.75) | -18.4 (2.82)
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.812, MMRM; Treatment Difference = -0.9, 95% CI 2-sided [-8.4 to 6.6] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.079, MMRM; Treatment Difference = -6.7, 95% CI 2-sided [-14.2 to 0.8] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.102, MMRM; Treatment Difference = -6.3, 95% CI 2-sided [-13.9 to 1.3] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]

8. Secondary Outcome: Change From Baseline in PhGA-PsA at Week 12
Description: The participants' overall disease status was assessed, taking into account signs, symptoms, and function, of all components of joint and skin affected at the time of the visit and this overall status was rated by the investigator using the PhGA-PsA VAS of 100 mm where 0 is 'very good, asymptomatic, and no limitation of normal activities' and 100 is 'very poor, very severe symptoms which are intolerable, and inability to carry out all normal activities'. A negative change from Baseline indicates improvement in symptoms.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 65 | 66 | 64 | 63
mm | -20.7 (2.66) | -29.6 (2.65) | -31.3 (2.65) | -31.6 (2.73)
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.016, MMRM; Treatment Difference = -8.9, 95% CI 2-sided [-16.2 to -1.7] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.004, MMRM; Treatment Difference = -10.6, 95% CI 2-sided [-17.8 to -3.4] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.003, MMRM; Treatment Difference = -10.9, 95% CI 2-sided [-18.2 to -3.6] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]

9. Secondary Outcome: Change From Baseline in HAQ-DI Total Score at Week 12
Description: The HAQ-DI consists of 20 questions referring to eight domains consisting of dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Each item is scored from 0 (without any difficulty) to 3 (unable to do). The worst score within each domain will be used as the domain score (i.e., if the score for one question is 1 and 2 for the other, then the worst score for the domain is 2). The HAQ-DI total score is calculated by dividing the sum of the domain scores by the number of non-missing domains. The total score indicates the patient's self-assessed level of functional ability and higher scores indicate worse functional ability. The HAQ-DI total score ranges from 0 to 3. A higher score indicates worse function and greater disability. A negative change from Baseline indicates improved function.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 66 | 66 | 64 | 63
score on a scale | -0.22 (0.053) | -0.29 (0.053) | -0.32 (0.053) | -0.28 (0.055)
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.357, MMRM; Treatment Difference = -0.07, 95% CI 2-sided [-0.21 to 0.08] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.195, MMRM; Treatment Difference = -0.10, 95% CI 2-sided [-0.24 to 0.05] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.467, MMRM; Treatment Difference = -0.05, 95% CI 2-sided [-0.20 to 0.09] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]

10. Secondary Outcome: Change From Baseline in Dactylitis Count (DC) at Week 12
Description: Tender score (0 = no tenderness, 1 = tender, 2 = tender and wince, 3 = tender and withdraw) is collected for Dactylitis Assessments on the Dactylitis Score Sheet that is used for calculation of total score. DC equals the number of tender fingers and toes (tender score >0). For participants with dactylitis status absent for all the fingers and toes, the DC is set as 0. The total score range of DC is from 0 to 60, higher scores indicate greater presence of dactylitis. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug. Overall number analyzed is the number of participants with dactylitis at Baseline and with available data.
Measure: Least Squares Mean (Standard Error); unit: dactylitis count
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 14 | 14 | 12 | 14
dactylitis count | -2.1 (0.39) | -0.8 (0.41) | -2.0 (0.47) | -1.9 (0.41)
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.031, MMRM; Treatment Difference = 1.3, 95% CI 2-sided [0.1 to 2.4] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.860, MMRM; Treatment Difference = 0.1, 95% CI 2-sided [-1.1 to 1.3] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.758, MMRM; Treatment Difference = 0.2, 95% CI 2-sided [-0.9 to 1.3] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]

11. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index (LEI) at Week 12
Description: Enthesitis is assessed using LEI. The enthesitis examination by LEI evaluates the presence or absence of pain by applying local pressure on 6 anatomical sites: medial femoral condyle (left and right), lateral epicondyle (left and right), and the achilles tendon insertion (left and right). Enthesitis at each site is scored as 0 (enthesitis absent) and 1 (enthesitis present). LEI is derived as the sum of the enthesitis score over the 6 sites, divided by the number of sites with non-missing score. The total score ranges from 0 to 6, higher scores indicate greater degree of enthesitis. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug. Overall number analyzed is the number of participants who had a baseline LEI score of ≥1 and with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 32 | 33 | 34 | 31
score on a scale | -0.9 (0.24) | -1.4 (0.24) | -1.6 (0.24) | -1.0 (0.25)
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.131, MMRM; Treatment Difference = -0.5, 95% CI 2-sided [-1.2 to 0.2] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.043, MMRM; Treatment Difference = -0.7, 95% CI 2-sided [-1.3 to 0.0] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.687, MMRM; Treatment Difference = -0.1, 95% CI 2-sided [-0.8 to 0.5] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]

12. Secondary Outcome: Percentage of Participants With Minimal Disease Activity (MDA) Response at Week 12
Description: MDA is a measure to indicate a state of minimal disease activity, and is a composite score of 7 domains. A participant is considered as having achieved the MDA if the participant fulfills at least 5 of the following 7 criteria: TJC 68 ≤1; SJC 66 ≤1; Psoriasis area and severity index (PASI) score ≤1 [The total score ranges from 0 (no disease) to 72 (maximal disease)] or body surface area (BSA) ≤3%; PGAAP ≤15 [using VAS on a scale of 0 (no pain) to 100 (serious pain)]; PGA-PsA ≤20 [using VAS on a scale of 0 (very well) to 100 (very poor)]; HAQ-DI score ≤0.5; LEI score ≤1. Percentages are rounded off to the nearest decimal.
Time Frame: Week 12
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 72 | 71 | 75 | 72
percentage of participants | 12.5 [4.9 to 20.1] | 18.3 [9.3 to 27.3] | 28.0 [17.8 to 38.2] | 29.2 [18.7 to 39.7]
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.349, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.6, 95% CI 2-sided [-6.1 to 17.4] — [estimate comment as in outcome 1, analysis 2]; Comparisons of MDA responder rates at Week 12 were made independently between each dose group and the placebo group using two-sided MH tests stratified on randomization stratification factors: prior treatment with biologics or non-traditional DMARDs and region
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.017, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.5, 95% CI 2-sided [2.8 to 28.3] — [estimate comment as in outcome 1, analysis 2]; [other analysis details as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.014, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.3, 95% CI 2-sided [3.3 to 29.3] — [estimate comment as in outcome 1, analysis 2]; [other analysis details as in outcome 12, analysis 1]

13. Secondary Outcome: Change From Baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) at Week 12
Description: The DAPSA score is a composite score and was calculated using: TJC68, SJC66, PGA-PsA, PGAAP, and hsCRP level (milligram per deciliter [mg/dL]). DAPSA scores 0-4 = remission, 5-14 = low disease activity, 15-28 = moderate disease activity, and >28 = high disease activity. The DAPSA score has a lower bound of 0 and has no upper bound. A higher DAPSA score indicated more active disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 64 | 64 | 63 | 62
score on a scale | -11.56 (1.948) | -15.30 (1.946) | -17.99 (1.943) | -16.79 (1.989)
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.167, MMRM; Treatment Difference = -3.73, 95% CI 2-sided [-9.04 to 1.57] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.018, MMRM; Treatment Difference = -6.43, 95% CI 2-sided [-11.73 to -1.13] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.056, MMRM; Treatment Difference = -5.23, 95% CI 2-sided [-10.59 to 0.13] — Point estimate and 95% CI were obtained from a MMRM model; [other analysis details as in outcome 4, analysis 1]

14. Secondary Outcome: Percentage of Participants Who Achieved PASI-75 Response at Week 12
Description: PASI-75 is assessed in participants with psoriasis involvement for ≥ 3% of the BSA at Baseline and assesses the extent of involvement and severity of psoriasis. To calculate the PASI, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). For PASI-75, the improvement threshold from baseline in PASI score is 75%. A higher score indicates more severe disease. Percentages are rounded off to the nearest decimal.
Time Frame: Week 12
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug. Overall number analyzed is the number of participants with psoriasis covering ≥ 3% of the BSA at Baseline and with available data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 39 | 39 | 46 | 46
percentage of participants | 15.4 [4.1 to 26.7] | 25.6 [11.9 to 39.3] | 28.3 [15.2 to 41.3] | 45.7 [31.3 to 60.0]
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.186, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.9, 95% CI 2-sided [-5.7 to 29.4] — [estimate comment as in outcome 1, analysis 2]; Comparisons of PASI-75 responder rates at Week 12 were made independently between each dose group and the placebo group using two-sided MH tests stratified on randomization stratification factors: prior treatment with biologics or non-traditional DMARDs and region
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.101, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.6, 95% CI 2-sided [-2.8 to 32.1] — [estimate comment as in outcome 1, analysis 2]; [other analysis details as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 29.0, 95% CI 2-sided [10.5 to 47.6] — [estimate comment as in outcome 1, analysis 2]; [other analysis details as in outcome 14, analysis 1]

15. Secondary Outcome: Percentage of Participants Who Achieved a Physician Global Assessment of Psoriasis (PhGA-PsO) of 0 or 1 and at Least a 2-point Improvement at Week 12
Description: PhGA-PsO responder is defined as participants 1) who had PhGA-PsO score of 0 or 1 at any given post-baseline visit; and 2) who had at least 2-point improvement from baseline. The PhGA-PsO is measured using a 0 to 4 scale with a 0 meaning clear or a 4 meaning severe. The proportion of participants achieving PhGA-PsO response at Week 12 was calculated and analyzed for participants with a score of at least 2 at baseline. Percentages are rounded off to the nearest decimal.
Time Frame: Week 12
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug. Overall number analyzed is the number of participants with PhGA-PSO ≥2 at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 57 | 54 | 63 | 58
percentage of participants | 15.8 [6.3 to 25.3] | 20.4 [9.6 to 31.1] | 20.6 [10.6 to 30.6] | 32.8 [20.7 to 44.8]
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 Low Dose; Test type: Superiority; p = 0.540, Cochran-Mantel-Haenszel; Risk Difference (RD) = 4.5, 95% CI 2-sided [-10.0 to 19.0] — [estimate comment as in outcome 1, analysis 2]; Comparisons of PhGA-PSO responder rates at Week 12 were made independently between each dose group and the placebo group using two-sided MH tests stratified on randomization stratification factors: prior treatment with biologics or non-traditional DMARDs and region
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 Medium Dose; Test type: Superiority; p = 0.466, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.2, 95% CI 2-sided [-8.8 to 19.3] — [estimate comment as in outcome 1, analysis 2]; [other analysis details as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 High Dose; Test type: Superiority; p = 0.034, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.3, 95% CI 2-sided [1.2 to 31.3] — [estimate comment as in outcome 1, analysis 2]; [other analysis details as in outcome 15, analysis 1]

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: Adverse Event(AE)=medical occurrence that does not necessarily have a causal relationship with this drug also including clinically meaningful findings in laboratory safety tests,vital signs,weight,and electrocardiogram(ECG).TEAEs=AEs occurring at time of or post study drug dosing until study end.SAE=any medical occurrence at any dose that resulted in death,was life-threatening,required inpatient hospitalization/prolongation of existing hospitalization,resulted in persistent or significant disability/incapacity,was a congenital abnormality/birth defect,an important medical event.AESIs included Common Terminology Criteria for Adverse Events(CTCAE)Grade≥2 cytopenia,CTCAE Grade≥3 elevation of creatine phosphokinase(CPK)[clinically significant or not]defined as CPK>5xupper limit of normal(ULN),infections,adverse events of abnormal liver function tests,adverse events of renal dysfunction,major adverse cardiovascular events,thromboembolic events,gastrointestinal perforation,and malignancies.
Time Frame: From first dose of study drug up to end of study (up to Week 16)
Population: Safety Analysis Set included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 72 | 71 | 75 | 72
Participants
  TEAEs | 39 | 42 | 45 | 56
  SAEs | 4 | 4 | 3 | 2
  AESIs | 19 | 33 | 22 | 38

17. Secondary Outcome: Plasma Concentration of NDI-034858
Description: Plasma concentration of NDI-034858 was measured in participants who received low, medium, or high doses of NDI-034858.
Time Frame: Pre-dose, 1 hour post-dose on Day 1 and Week 4, 4 hours post-dose at Week 4, Pre-dose at Week 8, and anytime at Week 12
Population: Pharmacokinetic (PK) Analysis Set included all participants in the Safety Analysis Set with at least one evaluable post-dose PK assessment. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
Number analyzed (Participants) | 71 | 75 | 72
nanograms per milliliter (ng/mL)
  Day 1: Pre-dose: number analyzed (Participants) | 66 | 75 | 71
  Day 1: Pre-dose | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  Day 1: 1 Hour: number analyzed (Participants) | 71 | 74 | 72
  Day 1: 1 Hour | 5.860 (7.251) | 25.43 (37.21) | 38.32 (59.74)
  Week 4: Pre-dose: number analyzed (Participants) | 67 | 66 | 65
  Week 4: Pre-dose | 25.26 (17.95) | 82.11 (74.46) | 187.5 (140.9)
  Week 4: 1 Hour: number analyzed (Participants) | 64 | 61 | 62
  Week 4: 1 Hour | 33.03 (24.05) | 112.8 (81.19) | 245.3 (184.6)
  Week 4: 4 Hours: number analyzed (Participants) | 64 | 61 | 61
  Week 4: 4 Hours | 46.68 (25.85) | 149.5 (90.56) | 370.1 (178.4)
  Week 8: Pre-dose: number analyzed (Participants) | 67 | 67 | 62
  Week 8: Pre-dose | 26.99 (21.00) | 78.29 (69.37) | 209.4 (182.0)
  Week 12: Any Time: number analyzed (Participants) | 61 | 61 | 58
  Week 12: Any Time | 24.85 (20.58) | 66.17 (51.81) | 178.2 (149.5)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study (up to Week 16)
Description: All-cause Mortality: all enrolled participants. SAEs and Other AEs: Safety Analysis Set included all randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | NDI-034858 Low Dose | NDI-034858 Medium Dose | NDI-034858 High Dose
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76 | 0/78 | 0/76
Serious Adverse Events (participants affected / at risk) | 4/72 | 4/71 | 3/75 | 2/72
Other Adverse Events (participants affected / at risk) | 13/72 | 19/71 | 27/75 | 35/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | NDI-034858 Low Dose (N=71) | NDI-034858 Medium Dose (N=75) | NDI-034858 High Dose (N=72)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | NDI-034858 Low Dose (N=71) | NDI-034858 Medium Dose (N=75) | NDI-034858 High Dose (N=72)
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 6
Blood creatine phosphokinase increased (Investigations) | 3 | 2 | 4 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 6
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 4
Headache (Nervous system disorders) | 3 | 2 | 6 | 4
Nasopharyngitis (Infections and infestations) | 3 | 6 | 7 | 7
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 6 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 8 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT05153148/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT05153148/SAP_001.pdf